CLINICAL TRIAL: NCT07043335
Title: Comparison of the Efficacy of Mesotherapy and Extracorporeal Shock Wave Therapy in Patients With Lateral Epicondylitis: A Prospective Randomised Controlled Trial
Brief Title: Comparison of the Efficacy of Mesotherapy and Extracorporeal Shock Wave Therapy in Patients With Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Gunay, MD, Specialist Physician, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMU-GETAT-KAEK/27.03.2024/04
Record Dates: First submitted 2024-12-19; First posted 2025-06-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: elbow pain; mesotherapy; lateral epicondylitis; extracorporeal shock wave therapy
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Mesotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Mesotherapy group) (Active Comparator): The intradermal mesotherapy will be applied to the painful points in the elbow using a 4 mm long, 30G needle with a point-by-point technique at a 90-degree angle. The injection volume per point will be 0.1 cc. Following this, a "nappage" technique with a 45-degree angle will be applied around the common extensor tendon.Mesotherapy solution will contain 1 cc 0.1% lidocaine, 1 cc pentoxifylline, 1 cc thiocolchicoside, 1 cc meloxicam 1⁄4 diluted with 0.9% physiological isotonic saline. Patients will receive a total of 5 sessions of mesotherapy, with one session every 7 days.
  Interventions: Procedure: Mesotherapy
- Group 2 (ESWT group) (Active Comparator): For patients in Group 2, Extracorporeal Shock Wave Therapy will be applied to the lateral epicondyle area at 10-15 Hz frequency, 1.5-2.5 bar energy density, and 2000 pulses. Patients will receive a total of 5 sessions of Extracorporeal Shock Wave Therapy (ESWT), with one session every 7 days.
  Interventions: Device: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — For patients in Group 2, Extracorporeal Shock Wave Therapy will be applied to the lateral epicondyle area at 10-15 Hz frequency, 1.5-2.5 bar energy density, and 2000 pulses. Patients will receive a total of 5 sessions of Extracorporeal Shock Wave Therapy (ESWT), with one session every 7 days.
  Arms: Group 2 (ESWT group)
Procedure: Mesotherapy — Intradermal mesotherapy involving lidocaine, pentoxifylline, meloxicam, and thiocolchicoside will be applied to painful elbow points using a 4 mm, 30G needle in a point-by-point technique at a 90° angle (0.1 cc per point). A nappage technique at a 45° angle will then be applied around the common extensor tendon. A total of five sessions will be administered, one every 7 days.
  Arms: Group 1 (Mesotherapy group)

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of mesotherapy in patients with lateral epicondylitis and to determine whether it is as effective as extracorporeal shock wave therapy (ESWT).

Is mesotherapy an effective method in patients with lateral epicondylitis?

Researchers will compare Mesotherapy to extracorporeal shock wave therapy (ESWT) in patient with Lateral epicondylitis.

Patients will be randomly assigned to either the Mesotherapy group or the ESWT group using a closed envelope method.

* Group 1 (Mesotherapy group): Patients will receive a total of 5 sessions of mesotherapy, with one session every 7 days.
* Group 2 (ESWT group): Patients will receive a total of 5 sessions of Extracorporeal Shock Wave Therapy (ESWT), with one session every 7 days.

Patients will be assessed at three time points: before treatment, 30 minutes after the completion of the treatment, and 12 weeks after the completion of the treatment

DETAILED DESCRIPTION:
This randomised-controlled single-blind prospective study was carried out at a Physical Medicine and Rehabilitation out-patient clinic. After approval by the Ethics Committee, all participants signed a written informed consent form. The research was conducted in accordance with the Helsinki Declaration.

Participants

The study will include individuals with lateral epicondylitis who are between the ages of 18 and 65 and have had elbow pain for at six weeks. Pain around the lateral epicondyle during resisted extension of wrist and fingers and tenderness over the lateral epicondyle were required for the diagnosis of lateral epicondylitis. Patients with the following exclusion criteria were not accepted into the study:

* Receiving an interventional injection in the elbow region within the last 3 months
* Receiving physical therapy in the last 3 months
* Receiving regular nonsteroidal anti-inflammatory drug (NSAID) treatment in the last 2 weeks
* History of fracture or surgery in the affected elbow region
* Chronic inflammatory diseases
* Acute infection
* History of malignancy
* Coagulation disorders
* Pregnancy
* Presence of a pacemaker or electronic implants
* Cervical radiculopathy and entrapment neuropathy
* Drug allergies
* BMI > 35

Demographic informations were recorded. Severity of elbow pain in activity were recorded according to Visual analogue Scale (VAS). Functional impairment were evaluated with The Patient-Rated Tennis Elbow Evaluation , Short-Form-Health-Survey-12 (SF-12 )

Following clinical assessment, patients were divided into two treatment groups randomly. Mesotherapy and Extracorporeal Shock wave Therapy . Exercise and resting wrist splints were recommended for all groups.

The first group received mesotherapy: For this group, a solution containing 1 cc each of lidocaine, pentoxifylline, thiocolchicoside, and meloxicam diluted ¼ with saline will be made. A 30 gauge, 4 mm mesotherapy injector will be used for the application. The lateral epicondyle will be the site of an intradermal injection. Of that amount, 2.5 cc will be applied point-by-point at intervals of 1-2 cm, and the remaining 2.5 cc will be applied using the napage method, 0.1 cc of solution were given with each injection.

Group 2 received Extracorporeal Shock Wave Therapy will be applied to the lateral epicondyle area at 10-15 Hz frequency, 1.5-2.5 bar energy density, and 2000 pulses. Patients will receive a total of 5 sessions of Extracorporeal Shock Wave Therapy (ESWT), with one session every 7 days.

All measures were conducted at baseline, after treatment, at 12 weeks follow-ups.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 65 years
* Pain and tenderness in the unilateral lateral epicondyle for ≥6 weeks
* Clinically diagnosed with Lateral Epicondylitis
* Patients without cognitive deficits who can follow verbal instructions Exclusion Criteria
* Receiving an interventional injection in the elbow region within the last 3 months
* Receiving physical therapy in the last 3 months
* Receiving regular nonsteroidal anti-inflammatory drug (NSAID) treatment in the last 2 weeks
* History of fracture or surgery in the affected elbow region
* Chronic inflammatory diseases
* Acute infection
* History of malignancy
* Coagulation disorders
* Pregnancy
* Presence of a pacemaker or electronic implants
* Cervical radiculopathy and entrapment neuropathy
* Drug allergies
* BMI > 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
VAS | All measures were conducted at baseline, at the end of treatment (Week 5), at 12th weeks follow-up
  Measurement of pain intensity using the Visual Analogue Scale (VAS). The VAS consists of a 10 cm line with endpoints representing 0 ("no pain") and 10 ("pain as bad as it could possibly be").
  Minimum score: 0
  Maximum score: 10
  Higher scores indicate worse pain.
Patient-Rated Tennis Elbow Evaluation | All measures were conducted at baseline, At the end of treatment (Week 5), at 12th weeks follow-ups
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis (tennis elbow). Scores range from 0 to 100, with higher scores indicating greater pain and disability.
SF-12 Health Survey | All measures were conducted at baseline,At the end of treatment (Week 5) , 12th weeks follow-ups
  A self-reported measure assessing health-related quality of life. Scores range from 0 to 100, with higher scores indicating better health status.

SECONDARY OUTCOMES:
Algometer Measurement of Pressure-Pain Threshold | All measures were conducted at baseline,At the end of treatment (Week 5) , at 12th weeks follow-ups.
  Measurement of pressure-pain threshold using an algometer device. Values are measured in kilopascals (kPa). Higher values indicate higher pain tolerance.
Hand Dynamometer for Grip Strength | All measures were conducted at baseline,At the end of treatment (Week 5) , at 12th weeks follow-ups.
  Measurement of grip strength using a hand dynamometer. Values are measured in kilograms (kg). Higher values indicate stronger grip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Haydarpasa Numune Research and Training Hospital, Istanbul, Uskudar 34668, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Mammucari M, Gatti A, Maggiori S, Sabato AF. Role of mesotherapy in musculoskeletal pain: opinions from the italian society of mesotherapy. Evid Based Complement Alternat Med. 2012;2012:436959. doi: 10.1155/2012/436959. Epub 2012 May 13. PMID 22654954
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22654954/